CLINICAL TRIAL: NCT03614728
Title: A Phase I/II Study to Investigate the Safety and Clinical Activity of GSK3326595 and Other Agents in Participants With Myelodysplastic Syndrome and Acute Myeloid Leukaemia
Brief Title: Study to Investigate the Safety and Clinical Activity of GSK3326595 and Other Agents to Treat Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial terminated due to internal review of clinical data in context of indication under investigation
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 208809
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Neoplasms
Keywords: Acute myeloid leukemia; Myelodysplastic syndrome; Chronic myelomonocytic leukemia; GSK3326595; 5-Azacitidine
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — GSK-3326595; Azacitidine

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, multi-part study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Participants receiving GSK3326595 (Experimental)
  Interventions: Drug: GSK3326595
- Part 2 Dose escalation : Participants receiving GSK3326595+5-Azacitidine (Experimental)
  Interventions: Drug: GSK3326595; Drug: 5-Azacitidine
- Part 2 Dose expansion: Participants receiving GSK3326595+5-Azacitidine (Experimental)
  Interventions: Drug: GSK3326595; Drug: 5-Azacitidine

INTERVENTIONS:
Drug: GSK3326595 — GSK3326595 will be administered.
Drug: 5-Azacitidine — 5-Azacitidine will be administered.
  Arms: Part 2 Dose escalation : Participants receiving GSK3326595+5-Azacitidine; Part 2 Dose expansion: Participants receiving GSK3326595+5-Azacitidine

SUMMARY:
This study will evaluate the safety, tolerability, and clinical activity of GSK3326595 in participants with relapsed and refractory MDS, chronic myelomonocytic leukemia (CMML), and AML. The study will be conducted in 2 parts: Part 1 will determine the clinical benefit rate (CBR) of GSK3326595 in monotherapy and Part 2 will be expanded to study GSK3326595 in combination with 5-Azacitidine which will be composed of a dose escalation phase followed by dose expansion cohort of GSK3326595.

ELIGIBILITY:
Inclusion Criteria:

* Males and females greater than or equal to (>=)18 years of age (at the time consent is obtained).
* Diagnosis of MDS, CMML or AML
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 or 2
* Adequate organ function
* A woman of childbearing potential (WOCBP) must have a negative highly sensitive serum pregnancy test within 7 days before the first dose of study intervention.

Exclusion Criteria:

* History of, or known, central nervous system (CNS) involvement
* Prior solid organ transplantation
* Known allergies, hypersensitivity, or intolerance to GSK3326595 or 5-Azacitidine or its excipient
* Prior therapy with any Protein arginine methyl transferase 5 (PRMT5) inhibitor
* History of a second malignancy, excluding non-melanoma skin cell cancer, within the last three years
* Active severe or uncontrolled infection
* History of optic nerve neuropathy or neuritis.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (6):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Watts J, Minden MD, Bachiashvili K, Brunner AM, Abedin S, Crossman T, Zajac M, Moroz V, Egger JL, Tarkar A, Kremer BE, Barbash O, Borthakur G. Phase I/II study of the clinical activity and safety of GSK3326595 in patients with myeloid neoplasms. Ther Adv Hematol. 2024 Sep 14;15:20406207241275376. doi: 10.1177/20406207241275376. eCollection 2024. PMID 39290981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study in participants with myeloid malignancies. Part 1 determined the clinical activity of GSK3326595 as monotherapy. Part 2 composed of a dose escalation and dose expansion cohorts to evaluate safety and clinical activity of GSK3326595 in combination with 5-Azacitidine
Pre-assignment Details: A total 30 participants were enrolled in Part 1. Part 2 was terminated early following a review of clinical data collected across the GSK3326595 clinical development program. Hence, no participants were enrolled in Part 2. The decision to terminate the study was not related to new safety concerns or to a change in the benefit risk profile of GSK3326595 .
Groups:
- Part 1: GSK3326595 400 mg: Participants received GSK3326595 400 milligram (mg), tablets, orally, once daily until progression, unacceptable toxicity, or withdrawal of consent during Part 1 of the study.
- Part 1: GSK3326595 300 mg: Participants received GSK3326595 300 mg, tablets, orally, once daily until progression, unacceptable toxicity, or withdrawal of consent during Part 1 of the study.
- Part 2-Dose Escalation: GSK3326595+5-Azacitidine: Participants were planned to receive GSK3326595 in combination with 5-Azacitidine in dose escalation cohort during Part 2 of the study.
- Part 2-Dose Expansion: GSK3326595+5-Azacitidine: Participants were planned to receive GSK3326595 in combination with 5-Azacitidine in dose expansion cohort during Part 2 of the study.
Period: Part 1 (Up to 30.8 Months)
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Started | 13 | 17 | 0 | 0
Completed | 12 | 16 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Part 2 (Up to 3 Years and 2 Months)
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Population consisted of all participants who received at least one dose of GSK3326595 as monotherapy or at least one dose of both combination drugs as combination treatment. Data was not collected in Part 2 of the study as no participant was enrolled in Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine | Total
Number analyzed (Participants) | 13 | 17 | 0 | 0 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (9.25) | 72.8 (9.61) |  |  | 71.7 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 |  |  | 7
  Male | 10 | 13 |  |  | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 0 |  |  | 3
  Asian - East Asian Heritage | 1 | 0 |  |  | 1
  White - Arabic/North African Heritage | 1 | 0 |  |  | 1
  White - White/Caucasian/European Heritage | 8 | 14 |  |  | 22
  Mixed Race | 0 | 1 |  |  | 1
  Unknown | 0 | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants achieving a complete remission (CR), complete marrow remission (mCR), partial remission (PR), stable disease (SD) lasting at least 8 weeks, or hematologic improvement (HI), per International Working Group (IWG) criteria, where CR=Bone marrow:<=5 percent(%) myeloblasts with normal maturation of all cell lines; PR=Bone marrow blasts decreased by >=50% over pre-treatment but still >5%; mCR=Bone marrow: <=5% myeloblasts and decrease by >=50% over pre-treatment; SD= Failure to achieve at least PR, but no evidence of progression >8 weeks; HI=Erythroid (E): hemoglobin increase of >1.5 grams per deciliter (g/dL), HI-Platelet: increase of >30,000/milliliter (mL) (starting with >20,000/mL) and increase from <20,000/mL to >20,000/mL by >100%; HI-Neutrophil: increase of >100% and >500/microliter. Percentage values are rounded off.
Time Frame: Up to 30.8 months
Population: All Treated Population consisted of all participants who received at least one dose of GSK3326595 as monotherapy or at least one dose of both combination drugs as combination treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Part 1: GSK3326595 400 mg: Participants received GSK3326595 400 mg, tablets, orally, once daily until progression, unacceptable toxicity, or withdrawal of consent during Part 1 of the study.
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Percentage of Participants | 15 [1.9 to 45.4] | 18 [3.8 to 43.4]

2. Primary Outcome: Part 2: Number of Participants With Non-serious Treatment-emergent Adverse Events (Non-STEAEs) and Serious Treatment Emergent Adverse Events (STEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement. Treatment emergent adverse event (TEAE) is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. Number of participants with non-STEAEs and STEAEs were planned to be assessed.
Time Frame: Up to 3 years and 2 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part 2: Number of Participants With AEs by Severity
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with AEs by severity were planned to be assessed.
Time Frame: Up to 3 years and 2 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part 2: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: An event is considered to be a DLT if the event occurs within the first 28 days of treatment meeting one of the following criteria of toxicity, Hematologic: Grade 4 or greater treatment-emergent neutropenia, anemia, or thrombocytopenia, lasting for >=14 days in the absence of Investigational Product, that cannot be attributed to underlying disease as described in National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4; Non-hematologic: Hepatic toxicity that meets Liver Stopping Criteria, Grade 3 nausea, vomiting or diarrhea that does not improve within 72 hours despite appropriate supportive treatments, Grade 4 or greater nausea, vomiting, or diarrhea of any duration, Any other Grade 3 or greater clinically significant non-hematologic toxicity; Other: Inability to receive all planned doses, dose interruption and Grade 2 or higher toxicity. Number of participants with DLTs were planned to be assessed.
Time Frame: Up to 28 days
Population: DLT Evaluable Population is defined as participants who received at least 75 percent (%) of the planned doses of GSK3326595 and all seven planned doses of 5-Azacitidine (Part 2) within the 28-day DLT observation period or those who have had a DLT. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Part 2: Number of Participants With AEs Leading to Dose Interruptions, Dose Reductions and Treatment Discontinuation Due to AEs
Description: Number of participants with AEs leading to dose interruptions, dose reductions and treatment discontinuation due to AEs were planned to be assessed.
Time Frame: Up to 3 years and 2 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part 1: Number of Participants With Common Non-STEAEs and STEAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. TEAEs which were not serious, were considered as non-STEAEs.
Time Frame: Up to 30.8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Participants
  Common non-STEAEs | 12 | 17
  STEAEs | 11 | 12

7. Secondary Outcome: Part 1: Number of Participants With AEs by Severity
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of each AE was reported during the study and was assigned a grade according to the NCI-CTCAE. AEs severity were graded as: Grade 1=mild; Grade 2=moderate; Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening consequences and Grade 5=death related to AE.
Time Frame: Up to 30.8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Participants
  Grade 1 | 0 | 0
  Grade 2 | 1 | 0
  Grade 3 | 0 | 6
  Grade 4 | 5 | 6
  Grade 5 | 7 | 5

8. Secondary Outcome: Part 1: Number of Participants With DLTs
Description: An event is considered to be a DLT if the event occurs within the first 28 days of treatment meeting one of the following criteria of toxicity, Hematologic: Grade 4 or greater treatment-emergent neutropenia, anemia, or thrombocytopenia, lasting for >=14 days in the absence of Investigational Product, that cannot be attributed to underlying disease as described in NCI-CTCAE version 4; Non-hematologic: Hepatic toxicity that meets Liver Stopping Criteria, Grade 3 nausea, vomiting or diarrhea that does not improve within 72 hours despite appropriate supportive treatments, Grade 4 or greater nausea, vomiting, or diarrhea of any duration, Any other Grade 3 or greater clinically significant non-hematologic toxicity; Other: Inability to receive all planned doses, dose interruption and Grade 2 or higher toxicity.
Time Frame: Up to 28 days
Population: DLT Evaluable Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 10 | 16
Participants | 0 | 0

9. Secondary Outcome: Part 1: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants achieving a CR, mCR, or PR, per IWG criteria, where CR=Bone marrow: <=5% myeloblasts with normal maturation of all cell lines; PR=Bone marrow blasts decreased by >=50% over pre-treatment but still >5%; mCR= Bone marrow: ≤ 5% myeloblasts and decrease by >=50% over pre-treatment. Percentage values are rounded off.
Time Frame: Up to 30.8 months
Population: All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Percentage of Participants | 0 [0.0 to 24.7] | 6 [0.1 to 28.7]

10. Secondary Outcome: Part 1: Progression Free Survival
Description: Progression free survival is defined as time from first dose to disease progression, as defined by IWG criteria, or death due to any cause, whichever occurs earlier. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Up to 30.8 months
Population: All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Months | 0.99 [0.95 to 2.53] | 0.99 [0.95 to 2.43]

11. Secondary Outcome: Part 1: Overall Survival
Description: Overall survival is defined as time from first dose to death due to any cause.
Time Frame: Up to 30.8 months
Population: All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Months | 2.69 [2.14 to 12.98] | 2.96 [1.28 to 15.24]

12. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: Day 1:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour), 24hours(+/-2hour) post-dose
Population: Pharmacokinetic (PK) Population consisted of all participants from the All Treated Population for whom a PK sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Nanogram per milliliter | 1322.8 (50) | 960.4 (61)

13. Secondary Outcome: Part 1: Cmax of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: Day 15:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour), 24hours(+/-2hour) post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 10 | 17
Nanogram per milliliter | 1125.4 (95) | 889.7 (38)

14. Secondary Outcome: Part 1: Time of Maximum Concentration Observed (Tmax) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Hours | 2.0000 [0.950 to 4.167] | 2.1667 [0.500 to 5.933]

15. Secondary Outcome: Part 1: Tmax of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 10 | 17
Hours | 2.9833 [0.083 to 5.833] | 2.9500 [0.483 to 4.067]

16. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t1/2) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 16
Hours | 5.0755 (45.248) | 6.7688 (52.542)

17. Secondary Outcome: Part 1: t1/2 of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 16
Hours | 6.2694 (47.757) | 6.8437 (67.132)

18. Secondary Outcome: Part 1: Area Under Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within Participant Across All Treatments (AUC[0-t]) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 17
Hours*nanogram per milliliter | 6667.4570 (56.989) | 5189.2734 (58.269)

19. Secondary Outcome: Part 1: AUC(0-t) of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 10 | 17
Hours*nanogram per milliliter | 5750.5167 (211.317) | 5651.2792 (49.506)

20. Secondary Outcome: Part 1: AUC From 0 Hours to the Time of Next Dosing (AUC[0-tau]) of GSK3326595
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 17
Hours*nanogram per milliliter | 8460 (65.8) | 5830 (45.0)

21. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC[0-inf]) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 16
Hours*nanogram per milliliter | 7128.4358 (54.648) | 6572.8527 (52.385)

22. Secondary Outcome: Part 1: AUC(0-inf) of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 16
Hours*nanogram per milliliter | 9202.5641 (70.085) | 6397.0840 (57.093)

23. Secondary Outcome: Part 1: Oral Clearance (CL/F) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 13 | 16
Liter per hour | 56.1133 (54.648) | 45.6423 (52.385)

24. Secondary Outcome: Part 1: CL/F of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 13
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 17
Liter per hour | 47.2832 (65.777) | 51.4710 (45.010)

25. Secondary Outcome: Part 1: Time Invariance Following Administration of GSK3326595
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595. Time invariance was calculated as the ratio of AUC(0-24) on Day 15 divided by AUC(0-infinity) on Day 1 for GSK3326595.
Time Frame: Days1and15:Pre-dose(within 1hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hour(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour),24hours(+/-2hour)post-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 16
Ratio | 1.3032 (46.471) | 0.9485 (57.938)

26. Secondary Outcome: Part 1: Accumulation Ratio Following Administration of GSK3326595
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595. Accumulation ratio was calculated as the ratio of AUC(0-24) on Day 15 divided by AUC(0-24) on Day 1 for GSK3326595.
Time Frame: as for outcome 25
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
Number analyzed (Participants) | 9 | 16
Ratio | 1.3814 (53.170) | 1.0774 (41.113)

27. Secondary Outcome: Part 2: Complete Remission (CR) Rate
Description: Complete remission rate is defined as percentage of participants achieving a CR per IWG criteria.
Time Frame: Up to 3 years and 2 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Part 2: Cmax of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Part 2: Cmax of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: Day 8:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour), 24hours(+/-2hour) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part 2: Cmax of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: Day 1:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Part 2: Cmax of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: Day 8:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Part 2: Tmax of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Part 2: Tmax of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Part 2: Tmax of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 30
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Part 2: Tmax of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part 2: t1/2 of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Part 2: t1/2 of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Part 2: t1/2 of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 30
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Part 2: t1/2 of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Part 2: AUC(0-t) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Part 2: AUC(0-t) of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Part 2: AUC(0-t) of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 30
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Part 2: AUC(0-t) of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Part 2: AUC(0-inf) of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Part 2: AUC(0-inf) of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Part 2: AUC(0-inf) of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 30
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Part 2: AUC(0-inf) of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Part 2: AUC(0-tau) Following Administration of GSK3326595
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Part 2: AUC(0-tau) Following Administration of 5-Azacitidine
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Part 2: CL/F of GSK3326595 Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 12
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Part 2: CL/F of GSK3326595 Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: as for outcome 29
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Part 2: CL/F of 5-Azacitidine Following Administration of Single Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 30
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Part 2: CL/F of 5-Azacitidine Following Administration of Repeat Dose
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 31
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Part 2: Time Invariance Following Administration of GSK3326595
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: Days 1 and 8:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour), 24hours(+/-2hour)post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Part 2: Time Invariance Following Administration of 5-Azacitidine
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: Days 1 and 8:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Part 2: Accumulation Ratio Following Administration of GSK3326595
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3326595.
Time Frame: Day 1 and 8:Pre-dose(within 1 hour prior to dosing),5minute(+/-2minute),30minute(+/-5minute),1hour(+/-5minute),2hours(+/-5minute),3hours(+/-5minute),4hours(+/-10minute),6hours(+/-10minute),8hours(+/-15minute),12hours(+/-2hour), 24hours(+/-2hour) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Part 2: Accumulation Ratio Following Administration of 5-Azacitidine
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of 5-Azacitidine.
Time Frame: as for outcome 55
Population: PK Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Part 2: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants achieving a CR, mCR, or PR, per IWG criteria.
Time Frame: Up to 3 years and 2 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2-Dose Escalation: GSK3326595+5-Azacitidine | Part 2-Dose Expansion: GSK3326595+5-Azacitidine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, common non-STEAEs and STEAEs were collected up to 30.8 months in Part 1 of the study
Description: All-cause mortality, common non-STEAEs and STEAEs were collected in Part A from All Treated Population. Data has been reported for only Part A and data were not collected for Part 2 as the study was terminated early and no participants were enrolled in Part 2 of the study.
Arm/Group | Part 1: GSK3326595 400 mg | Part 1: GSK3326595 300 mg
All-Cause Mortality (participants affected / at risk) | 11/13 | 14/17
Serious Adverse Events (participants affected / at risk) | 11/13 | 12/17
Other Adverse Events (participants affected / at risk) | 12/13 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GSK3326595 400 mg (N=13) | Part 1: GSK3326595 300 mg (N=17)
Sepsis (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 0
Actinomycosis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Asthenia (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GSK3326595 400 mg (N=13) | Part 1: GSK3326595 300 mg (N=17)
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Oral disorder (Gastrointestinal disorders) | 2 | 0
Rectal lesion (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal discomfort (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 4 | 8
Neutrophil count decreased (Investigations) | 2 | 6
International normalised ratio increased (Investigations) | 4 | 3
Blood creatinine increased (Investigations) | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Prothrombin time prolonged (Investigations) | 1 | 2
Troponin T increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 7
Headache (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 2 | 3
Balance disorder (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 7 | 6
Oedema peripheral (General disorders) | 5 | 2
Chills (General disorders) | 2 | 2
Pyrexia (General disorders) | 4 | 0
Asthenia (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nodular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Micturition frequency decreased (Renal and urinary disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03614728/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03614728/SAP_001.pdf